CLINICAL TRIAL: NCT01473303
Title: Phase IB/Randomized Phase II Study of Folfirinox Plus AMG-479 (Ganitumab) or Placebo in Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Brief Title: Combination Chemotherapy With or Without Ganitumab in Treating Patients With Previously Untreated Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: CALGB 81003 closed about a week after it was activated because of withdrawal of support. No patients were registered on this study.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-81003; CALGB-81003; CDR0000716301 (Registry Identifier: NCI Physician Reference Desk)
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Cancer
Keywords: stage IV pancreatic cancer; duct cell adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ganitumab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

ARMS (2):
- Arm I (Experimental): Patients receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 48 hours beginning on day 2 (mFOLFIRINOX) and ganitumab IV over 30-60 minutes on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ganitumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin
- Arm II (Experimental): Patients receive mFOLFIRINOX as in arm I and placebo IV over 30-60 minutes on day 1.
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin; Other: placebo; Other: questionnaire administration

INTERVENTIONS:
Biological: ganitumab — Given IV
  Arms: Arm I
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV
Drug: oxaliplatin — Given IV
Other: placebo — Given IV
  Arms: Arm II
Other: questionnaire administration — Completed on paper
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin calcium, irinotecan hydrochloride, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as ganitumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. It is not yet known whether giving more than one drug (combination chemotherapy) is more effective with or without ganitumab in treating patients with pancreatic cancer.

PURPOSE: This phase I/II trial is studying the best dose of combination chemotherapy and ganitumab and how well combination chemotherapy with or without ganitumab works in treating patients with previously untreated metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety and determine the maximally tolerated dose (MTD) of modified FOLFIRINOX (mFOLFIRINOX) and ganitumab in patients with previously untreated, metastatic pancreatic adenocarcinoma. (phase I)
* To compare overall survival of patients with previously untreated, metastatic pancreatic adenocarcinoma who receive mFOLFIRINOX plus ganitumab versus mFOLFIRINOX plus placebo. (phase II)
* To assess the convergent validity of each selected PRO-CTCAE item by comparing each item at baseline between patients with ECOG performance status (PS) 0 vs 1. (phase II)

Secondary

* To compare objective response rate, duration of response, and progression-free survival of patients with previously untreated, metastatic pancreatic adenocarcinoma who receive mFOLFIRINOX plus ganitumab versus mFOLFIRINOX plus placebo.
* To compare treatment-related toxicity in patients with previously untreated, metastatic pancreatic adenocarcinoma who receive mFOLFIRINOX plus ganitumab versus mFOLFIRINOX plus placebo.
* To assess the responsiveness (sensitivity to change) of Patient-Reported Outcomes (PRO)-CTCAE by comparing change scores within groups of patients as defined by changes in ECOG PS at post-baseline administrations. (phase II)
* To compare the maximum post-baseline score for each PRO-CTCAE item per patient between arms in the randomized phase II component of the study. (exploratory).

OUTLINE: This is a dose-escalation, phase IB study followed by a randomized phase II study. Patients in the phase II study are stratified according to ECOG performance status of 0 versus 1.

* Phase IB: Patients receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 48 hours beginning on day 2 (mFOLFIRINOX). After cohort 0, subsequent patients also receive ganitumab IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients are randomized to 1 of 2 treatment arms:

  * Arm I: Patients receive mFOLFIRINOX as in Phase IB and ganitumab IV over 30-60 minutes on day 1.
  * Arm II: Patients receive mFOLFIRINOX as in Phase IB and placebo IV over 30-60 minutes on day 1.

In both arms, treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Patients randomized in the phase II component of the study may complete 16 Patient-Reported Outcomes (PRO)-CTCAE items (measuring 8 symptoms) on paper on day 1 of all odd-numbered courses (i.e., courses 1, 3, 5, etc.).

Tumor tissue and blood samples may be collected for correlative studies.

After completion of study therapy, patients are followed every 3 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma
* Metastatic disease to distant sites, as documented by CT scan or MRI

  * Patients with locally advanced disease are NOT eligible
* At least one site of disease measurable by RECIST 1.1 criteria; defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 2 cm with conventional techniques or as ≥ 1 cm with spiral CT scan
* No known CNS metastases or carcinomatous meningitis, as determined by physical examination and/or imaging studies
* No suspected Gilbert syndrome or known homozygosity for the UGT1A1*28 allele (UGT1A1 genotyping is not required for enrollment on this study; however, patients known to be homozygous for the UGT1A1*28 allele are excluded)

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* Neutrophils ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN
* INR ≤ 1.5
* Blood glucose level ≤ 160 mg/dL

  * Patients with non-fasting blood glucose > 160 mg/dL must have a fasting blood glucose ≤ 160 mg/dL to be eligible
  * Patients with diabetes mellitus are allowed at the discretion of the treating investigator, if blood sugars are felt to be under appropriate control
* Not pregnant or nursing
* Negative serum or urine pregnancy test
* No malignancy (other than non-melanoma skin cancer or carcinoma in situ of the cervix) diagnosed within the past 3 years or any currently active malignancy

  * A malignancy is considered not "active" if all anti-cancer therapies were completed > 3 years before enrollment and there is no current evidence of persistent disease
* No neurosensory or neuromotor toxicity ≥ grade 2
* No known allergy to platinum compounds or E. coli-derived products (e.g., filgrastim, humulin, insulin, or L-asparaginase)
* No colonic or small bowel disorders with uncontrolled symptoms at baseline (for example, > 3 watery or soft stools daily in patients without colostomy or ileostomy)

  * Patients with colostomy or ileostomy can be enrolled at the discretion of the investigator
* No history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within 6 months of registration
* No HIV-positive patients with a prior history of AIDS-defining illness

  * No HIV-positive patients with a CD4 count of < 450 cells/mm³ at any point prior to study
  * Anti-retroviral therapy must be discontinued during study treatment
* No known positivity for chronic infection with B virus (HBV)

PRIOR CONCURRENT THERAPY:

* Prior treatment with chemotherapy or radiotherapy for resected, locally advanced or metastatic pancreatic cancer is NOT allowed
* No prior treatment with inhibitors of the insulin-like growth factor 1 receptor
* No prior treatment with radiotherapy to greater than 25% of bone marrow
* Palliative radiation therapy may NOT be administered while a subject is on the study
* No major surgery within 4 weeks of the start of study treatment

  * Patients must have recovered from the side effects of any major surgery at the start of study treatment
  * Major surgery is defined as those surgeries that require general anesthesia

    * Insertion of a vascular access device or endobiliary stent is NOT considered major surgery
* No percutaneous biliary drain (endobiliary stents are allowed)
* Warfarin for INR goal > 1.5 is prohibited

  * Patients on warfarin with INR goal of ≤ 1.5 are eligible
* Hormones or other chemotherapeutic agents may NOT be administered except for steroids given for adrenal failure; hormones administered for non-disease-related conditions (e.g., insulin for diabetes); and intermittent use of dexamethasone as an antiemetic or for the prevention or treatment of ganitumab infusion reactions
* Patients receiving anti-retroviral therapy must discontinue such therapy while receiving study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (phase I)
Maximum-tolerated dose (phase I)
Overall survival (phase II)
Convergent validity of each selected PRO-CTCAE item (phase II)

SECONDARY OUTCOMES:
Objective response rate and duration of response between the mFOLFIRINOX plus ganitumab and the mFOLFIRINOX plus placebo arms (phase II)
Progression-free survival (phase II)
Responsiveness (sensitivity to change) of PRO-CTCAE (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Brain Wolpin, MD, Principal Investigator — Dana-Farber Cancer Institute